CLINICAL TRIAL: NCT06028854
Title: Association Between Preoperative Blood Characteristics and Mortality in Abdominal Emergency Surgeries
Brief Title: Blood Characteristics and Abdominal Emergency Surgery
Status: Suspended | Type: Observational
Why Stopped: The study was suspended because of difficulties in recruiting participants within the expected timeframe.
Sponsor: University of Chile (Other)
Responsible Party: Sponsor
Other Study IDs: OAIC 1337/23
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Surgical Wound
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- High Neutrophil count: Patients with high neutrophil count in their preoperative complete blood count
- Low Neutrophil count: Patients with low neutrophil count in their preoperative complete blood count

SUMMARY:
After surgical tissue damage, cellular blood components are involved in tissue repair processes, yet their preoperative characteristics are not considered in routine clinical practice.

DETAILED DESCRIPTION:
Surgical injuries initiate the recruitment of cellular blood components for tissue repair. Baseline inflammation levels and cellular response to tissue damage are absent from perioperative management algorithms despite their importance in regeneration. This project seeks to examine patients preoperative parameters before surgery and evaluate if there is a correlation with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years of age at surgery.
* Patients with acute intra-abdominal pathology requiring emergency surgery.
* A complete blood count was performed in the emergency department of our center within 24 hours before surgery.

Exclusion Criteria:

* Patients who are users of anticoagulation before admission for any reason
* Patients who have had previous hospitalization or surgery in the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acute intrabdominal pathology who requires surgery in the next 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Death | 1 year
  The number of deceased patients.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Maldonado, Study Chair — Hospital Clinico de la Universidad de Chile
Locations (2):
- Chile (2):
  - Hospital Clínico de la Universidad de Chile, Independencia, Santiago Metropolitan
  - Hospital Clínico Universidad de Chile, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: No